CLINICAL TRIAL: NCT03386513
Title: A Phase 1/2, Multi-center, Open-label Study of IMGN632 Monotherapy Administered Intravenously in Patients With CD123-positive Acute Myeloid Leukemia and Other CD123-positive Hematologic Malignancies
Brief Title: Study of IMGN632 in Patients With Untreated BPDCN and Relapsed/Refractory BPDCN
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMGN632-0801; 2024-514195-40-00 (EU CTIS Number)
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Blastic Plasmacytoid Dendritic Cell Neoplasm; Myeloproliferative Neoplasm
Keywords: Antibody Drug Conjugate; Other Hematologic Malignancies; Myeloproliferative Neoplasms; CD123; MDS; Relapsed, Refractory; Acute Lymphocytic Leukaemia; Blastic Plasmacytoid Dendritic Cell Neoplasm; Acute Myeloid Leukemia
MeSH Terms: conditions — Blastic Plasmacytoid Dendritic Cell Neoplasm; Myeloproliferative Disorders; Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Escalation and Expansion (Experimental): Escalation: IMGN632 was administered by IV on 2 different schedules for participants with relapsed/refractory AML, ALL, or BPDCN.
  Expansion: IMGN632 was administered by IV:
  * Cohort 1: Relapsed or refractory BPDCN participants who have received 1-3 prior systemic therapies (incl. tagraxofusp-erzs and/or any other systemic therapy deemed appropriate for the treatment of BPDCN)
  * Cohort 2: Relapsed AML
  * Cohort 3: Relapsed or refractory ALL
  * Cohort 4: Other relapsed or refractory hematologic malignancies
  * Cohort 5: Relapsed or refractory AML at alternate dose or schedule
  * Cohort 6: Pivotal cohort for frontline BPDCN participants who have not received prior systemic therapy and participants with frontline BPDCN who have prior or concomitant hematologic malignancy (PCHM) and have not received prior systemic therapy.
  Interventions: Drug: IMGN632

INTERVENTIONS:
Drug: IMGN632 — CD123-targeted ADC

SUMMARY:
This is an open-label, multi-center, Phase 1/2 study to determine the MTD and assess the safety, tolerability, PK, immunogenicity, and anti-leukemia activity of IMGN632 when administered as monotherapy to patients with CD123+ disease.

DETAILED DESCRIPTION:
IMGN632 is administered by IV on Day 1 of each cycle, with cycles repeating every 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Disease Characteristics:

   a. Confirmation of CD123 positivity by flow cytometry or IHC. Participants who received prior CD123-targeting agents will be allowed as long as the blasts still have detectable CD123 expression.
2. Expansion inclusion:

   * Cohort 1 - Participants with relapsed or refractory blastic plasmacytoid dendritic cell neoplasm (BPDCN) with 1-3 prior lines of therapy
   * Cohort 2 - Participants with relapsed AML
   * Cohort 3 - Participants with relapsed relapsed or refractory ALL (including any subtypes: B-cell, T-cell, Ph+ and Ph-)
   * Cohort 4 - Participants with relapsed or refractory other hematologic malignancies not included in the cohorts above (eg, high risk/very high-risk MDS, MPN, CMML, BP-CML).
   * Cohort 5 - Participants with relapsed relapsed or refractory (to nonintense therapies) CD123+ AML.
   * Cohort 6 - Participants with frontline de novo BPDCN at screening who have not received prior systemic therapy and participants with frontline BPDCN who have PCHM and have not received prior systemic therapy.

Note: Participants in Cohort 6 may have received local therapy (radiotherapy, surgical excision, photodynamic therapy). Eligible participants must have a recurrence or progression in the field of local therapy OR disease outside the field of local therapy.

Exclusion Criteria:

1. Participants who, in the judgment of their treating physician, have appropriate standard of care therapies will be excluded from Cohorts 1 through 5.
2. Frontline BPDCN participants with central nervous system (CNS) disease will be excluded. A lumbar puncture must be performed during the 28-day screening period, prior to drug administration. Relapsed or refractory BPDCN participants with a known history of CNS disease must have been treated locally, have at least 1 lumbar puncture with no evidence of CNS disease, and must be clinically stable prior to first dose. Concurrent therapy for CNS prophylaxis or continuation of therapy for controlled CNS disease is permitted with the approval of the Sponsor.
3. Participants with a history of veno-occlusive disease (sinusoidal obstruction syndrome) of the liver.
4. Participants with a history of Grade 4 capillary leak syndrome, or non-cardiac Grade 4 edema are ineligible, eg, related to tagraxofusp-erzs or other etiology.
5. Interval from prior cancer therapy: 1. For frontline BPDCN participants with prior local therapy (eg, radiotherapy), participants must not have received treatment within 14 days prior to drug administration on this study. 2. Relapsed or refractory BPDCN participants must not have received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal, biologic, or any investigational agents within 14 days prior to drug administration on this study. Participants must have recovered to baseline from all acute toxicity from this prior therapy.

Note: the exception that participants who have received a checkpoint inhibitor must not have received that therapy within 28 days prior to drug administration on this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
To assess the rate of composite CR in BPDCN patients | 21-day cycle
  CR+clinical CR [CRc]

SECONDARY OUTCOMES:
To assess the duration of CR (DOCR) for patients with CR or CRc | Up to 24 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | Up to 24 months
To assess the rate of CR+CRc+CRh | Up to 24 months
To assess the duration of CR+CRc+CRh | Up to 24 months
To assess ORR: CR+CRc+CRh+CRi+PR | Up to 24 months
To assess the duration of overall response | Up to 24 months
To assess OS | Up to 24 months
To assess the percent of BPDCN patients able to bridge to stem cell transplant in the frontline and relapsed/refractory populations separately | Up to 24 months
To characterize the PK of IMGN632, total antibody, and FGN849 (the active catabolite) | Up to 24 months
To evaluate the potential immunogenicity of IMGN632 | Up to 24 months
  ADA
To assess transfusion independence | Up to 24 months
  Conversion rate to independence of red blood cell (RBC) and platelet transfusion relative to baseline

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (28):
- United States (15):
  - Banner Health MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope Medical Center, Duarte, California
  - UCLA, Los Angeles, California
  - Stanford, Stanford, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Novant Health Cancer Institute Hematology, Charlotte, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Novant Health Cancer Institute Hematology - Forsyth, Winston-Salem, North Carolina
  - Baylor Scott & White University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center/Seattle Cancer Care Alliance, Seattle, Washington
- France (5):
  - Recherche Clinique-Hématologie, Amiens
  - CHU de Besancon, Hopital Jean Minjoz, Besançon
  - Institut Paoli Calmettes (Marseille), Marseille
  - Hôpital St Antoine, Paris
  - CHU Bordeaux Hôpital Haut-Lévêque, Pessac
- Germany (2):
  - University Hospital of Cologne, Cologne
  - University Hospital of Leipzig, Leipzig
- Italy (4):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola Malpighi, Bologna
  - Instituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Instituto Europeo di Oncologia, Milan
  - Azienda ospedaliera Santa Maria della Misericordia, Perugia
- Hospital Universitari I Politècnic La Fe, Valencia, Spain
- Churchill Hospital - Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daver NG, Montesinos P, DeAngelo DJ, Wang ES, Papadantonakis N, Todisco E, Sweet KL, Pemmaraju N, Lane AA, Torres-Minana L, Thompson JE, Konopleva MY, Sloss CM, Watkins K, Bedse G, Du Y, Malcolm KE, Zweidler-McKay PA, Kantarjian HM. Pivekimab sunirine (IMGN632), a novel CD123-targeting antibody-drug conjugate, in relapsed or refractory acute myeloid leukaemia: a phase 1/2 study. Lancet Oncol. 2024 Mar;25(3):388-399. doi: 10.1016/S1470-2045(23)00674-5. PMID 38423051